CLINICAL TRIAL: NCT07126561
Title: Phase II Open Label Trial of Trastuzumab Deruxtecan (Enhertu, DS-8210) in HER2 Positive Newly Diagnosed Metastatic Esophageal, Gastric, GEJ Cancer Patients With an ECOG Performance Status of 2
Brief Title: Trastuzumab Deruxtecan to Treat HER2 + Newly Diagnosed Metastatic GI Cancers
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB25-1217
Record Dates: First submitted 2025-08-11; First posted 2025-08-17 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-07

CONDITIONS: HER2 Positive Newly Diagnosed Metastatic Esophageal, Gastric, GEJ Cancer Patients With an ECOG Performance Status of 2
Keywords: HER2; TRASTUZUMAB; DERUXTECAN; METASTATIC; CANCER; ESOPHAGEAL; GASTRIC; GEJ
MeSH Terms: conditions — Neoplasm Metastasis; Neoplasms | interventions — trastuzumab deruxtecan

STUDY DESIGN:
Intervention Model Description: Simon's two-stage optimal design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- multicenter single-arm phase II open label trial of Trastuzumab Deruxtecan (Enhertu, DS-8210). (Experimental)
  Interventions: Drug: Trastuzumab Deruxtecan

INTERVENTIONS:
Drug: Trastuzumab Deruxtecan — Do not substitute trastuzumab deruxtecan with trastuzumab or ado-trastuzumab emtansine. Do not administer as an intravenous push or bolus. Trastuzumab deruxtecan is not compatible with sodium chloride 0.9% solution for infusion. During treatment, patients should be observed for infusion-related reactions (IRRs). For additional information on the management of IRRs

SUMMARY:
Purpose: This clinical trial is designed to evaluate the safety and effectiveness of Trastuzumab Deruxtecan for patients with HER2 Positive Newly Diagnosed Metastatic Esophageal, Gastric, GEJ Cancer. The goal is to determine how well this treatment works and to identify any potential side effects.

Who Can Participate: We are looking for Participants with histologically confirmed HER2 positive locally advanced unresectable and/or metastatic esophageal, gastric or GEJ adenocarcinoma with an ECOG PS of 2 and measurable disease according to RECIST 1.1 within 42 days prior to registration. Participants will be carefully screened to ensure they meet the study requirements.

What to Expect: Participants will undergo 6.4mg/kg, IV infusion of Trastuzumab deruxtucan over the course of the study. They will receive detailed information about the study and will have the opportunity to ask questions before deciding to participate. Informed consent will be obtained to ensure that participants understand the study's purpose, procedures, risks, and benefits.

Safety Monitoring: The health and safety of participants are our top priority. An Independent Data and Safety Monitoring Committee (DSMC) will regularly review the study data to ensure participant safety and to monitor for any adverse events. Any serious side effects will be reported and addressed promptly.

Benefits and Risks: While the study aims to provide potential benefits, such as improved treatment options for HER2 Positive Newly Diagnosed Metastatic Esophageal, Gastric, GEJ Cancer there may also be risks involved. Participants will be informed of all possible risks before enrolling in the study.

Confidentiality: All personal information will be kept confidential, and data will be used only for research purposes.

Contact Information: For more information about this study, please contact PhaseIICRA@medicine.bsd.uchicago.edu

ELIGIBILITY:
Inclusion Criteria:

* 1.1.1 Participants must agree to provide written informed consent and HIPAA authorization for release of personal health information prior to registration.

NOTE: HIPAA authorization may be included in the informed consent or obtained separately.

1.1.2 Participants must be ≥ 18 years of age at the time of consent.

1.1.3 Participants must have histologically confirmed locally advanced unresectable and/or metastatic esophageal, gastric or GEJ adenocarcinoma per AJCC, 8th edition.

1.1.4 Participants must have measurable disease according to RECIST 1.1 within 42 days prior to registration.

1.1.5 Participants must have an ECOG PS of Grade 2 within 28 days prior to registration.

1.1.6 Participants must NOT be candidates for combination therapy per treating provider judgement.

1.1.7 Participants must have HER2 protein overexpression or HER2 gene amplification in tumor tissue (preferred on tumor tissue biopsy if available) or liquid biopsy. (Note: HER2 levels considered positive Score 3+ on IHC, Score of 2+ with positive results of FISH)

1.1.8 Prior definitive chemoradiation therapy for localized disease, systemic therapy including immunotherapy in the adjuvant setting is allowed.

1.1.9 Prior cancer treatment in the adjuvant setting must be completed at least 3 months prior to registration and the participant must have recovered from all reversible acute toxic effects of the regimen (other than alopecia) to Grade ≤ 1 or baseline.

1.1.10 Participants must demonstrate adequate organ and bone marrow function within 28 days before registration as described in the table below. Organ and bone marrow function criteria must also be met when laboratory tests are repeated within 3 days before Cycle 1 Day 1.

1.1.1 Females of childbearing potential must have a negative serum pregnancy test within 7 days prior to registration. A negative result for serum pregnancy test (test must have a sensitivity of at least 25 mIU/mL) must be available at the screening visit and urine beta-human chorionic gonadotropin (β-HCG) pregnancy test prior to each administration of IMP.

Women of childbearing potential are defined as those who are not surgically sterile (i.e. underwent bilateral salpingectomy, bilateral oophorectomy, or complete hysterectomy) or post-menopausal. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause.

1.1.2 Females of childbearing potential who are sexually active with a male able to father a child must be willing to abstain from penile-vaginal intercourse or must use at least one highly effective method of contraception from the time of first exposure to study intervention until 7 months after the final dose. They must also refrain from breastfeeding or donating ova /retrieving ova for their own use for the same time period.

1.1.3 Males able to father a child who are sexually active with female of childbearing potential must be willing to abstain from penile-vaginal intercourse or must use at least one highly effective method of contraception from the time of first exposure to study intervention until 4 months after the final dose. They must also refrain from freezing or donating sperm during the same time period.

1.1.4 All participants must be able to understand and comply with study procedures for the entire length of the study, as determined by the enrolling physician or protocol designee.

Exclusion Criteria:

* 1.1.1 Prior systemic therapy in the metastatic setting is not allowed, including no prior HER2-directed therapy. However, prior palliative radiation therapy is allowed.

1.1.2 Participants who are eligible for combination therapy are excluded.

1.1.3 Participants who are mismatch repair (MMR) deficient and/or MSI High as determined by institutional standards are not eligible for this study.

1.1.4 Participants who have an LVEF <50% within 28 days before first exposure to study drug are not eligible for this study.

1.1.5 Participants who have unresolved toxicities from previous anticancer therapy, defined as toxicities (other than alopecia) not yet resolved to Grade ≤1 or baseline are excluded.

NOTE: Participants may be enrolled with chronic, stable Grade 2 toxicities (defined as no worsening to >Grade 2 for at least 3 months prior to first exposure to study intervention and managed with standard of care treatment) that the investigator deems related to previous anticancer therapy, including:

* Chemotherapy-induced neuropathy
* Fatigue
* Residual toxicities from prior immuno-oncology treatment: Grade 1 or Grade 2 endocrinopathies which may include:

  1. Hypothyroidism/hyperthyroidism
  2. Type 1 diabetes
  3. Hyperglycemia
  4. Adrenal insufficiency
  5. Adrenalitis
  6. Skin hypopigmentation (vitiligo)

     1.1.6 Participants with an active primary immunodeficiency, known uncontrolled active human immunodeficiency virus (HIV) infection, or active hepatitis B (HBV) or C (HCV) virus infection are excluded. Note: Hepatitis B/C serology is required; HIV testing is not required unless required by local policy.
* NOTE: Participants with past or resolved HBV infection are eligible only if they meet all of the following criteria:

  * HBsAg (-) (for > 6 months off anti-viral treatment);
  * Anti-HBc (+) (IgG or total Ig);
  * HBV DNA undetectable;
  * Liver architecture normal (absence of any liver pathology including absence of cirrhosis or fibrosis on prior imaging or biopsy;
  * Absence of HCV co-infection or history of HCV co-infection;
  * Access to a local Hepatitis B expert during and after the study;

Those participants must be closely monitored for HBV reactivation. Further instructions for monitoring and management of participants at risk of Hepatitis B reactivation (those with HBsAg (-), anti-HBc (+) (IgG or total Ig) serology) are provided in Appendix I.

• NOTE: Participants positive for HCV antibody are eligible only if polymerase chain reaction is negative for HCV RNA.

1.1.7 Participants with a medical history of myocardial infarction (MI) within 6 months before study registration or symptomatic congestive heart failure (New York Heart Association Class II to IV) are not eligible. Participants with troponin levels above ULN at screening, and without any myocardial related symptoms, should have a cardiologic consultation before enrollment to rule out MI.

1.1.8 Participants with a history of (non-infectious) ILD/pneumonitis that required steroids, has current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at screening.

1.1.9 Participants with a history of any of the following lung criteria are excluded:

* Lung-specific intercurrent clinically significant illnesses including, but not limited to, any underlying pulmonary disorder (e.g., pulmonary emboli within three months of registration, severe asthma, severe chronic obstructive pulmonary disorder, restrictive lung disease, pleural effusion, etc.)
* Any autoimmune, connective tissue or inflammatory disorders, including Rheumatoid arthritis, Sjogren's, and sarcoidosis, where there is documented, or a suspicion of pulmonary involvement at the time of screening. Full details of the disorder should be recorded in the eCRF for participants who are included in the study.
* Prior pneumonectomy (complete),

1.1.10 Participants who have spinal cord compression or clinically active central nervous system metastases, defined as untreated and symptomatic, or requiring therapy with corticosteroids or anticonvulsants to control associated symptoms are not eligible. Participants with clinically inactive brain metastases may be included in the study. Participants with treated brain metastases that are no longer symptomatic and who require no treatment with corticosteroids or anticonvulsants may be included in the study if they have recovered from the acute toxic effect of radiotherapy. A minimum of 2 weeks must have elapsed between the end of whole brain radiotherapy and study registration.

1.1.11 Participants with uncontrolled infection requiring IV antibiotics, antivirals, or antifungals.

1.1.12 Participants with a prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of the investigational regimen, per treating physician discretion, are not eligible for this trial.

1.1.13 Participants who have received treatment with any investigational anti-cancer drug within 2 weeks prior to registration are excluded.

Washout periods for other therapies are listed below:

Treatment Minimum Washout Chloroquine/Hydroxychloroquine ≥ 14 days Radiation Therapy including palliative stereotactic radiation therapy to chest ≥ 4 weeks Palliative stereotactic radiation therapy to other anatomic areas including whole brain radiation ≥ 2 weeks

1.1.14 Participants who have received live, attenuated vaccine (mRNA and replication deficient adenoviral vaccines are not considered attenuated live vaccines) within 30 days prior to study registration are excluded. NOTE: Participants, if enrolled, should not receive live vaccine during the study and up to 30 days after the last dose of study intervention.

1.1.15 Participant has substance abuse or any other medical conditions such as clinically significant cardiac or psychological conditions, that may, in the opinion of the investigator, interfere with the subject's participation in the clinical study or evaluation of the clinical study results.

1.1.16 Participant has Corrected QT interval (QTcF) prolongation to > 470 msec (females) or >450 msec (males) based on average of the screening triplicate12-lead ECG.

1.1.17 Participant has a known allergy or hypersensitivity to study treatment or any of the study drug excipients.

1.1.18 Participant has a history of severe hypersensitivity reactions to other monoclonal antibodies.

1.1.19 Participant has multiple primary malignancies within 3 years, with the exception of: adequately resected non-melanoma skin cancer, curatively treated in-situ disease. other solid tumors curatively treated

1.1.20 Participant has a pleural effusion, ascites or pericardial effusion that requires drainage, peritoneal shunt, or Cell-free and Concentrated Ascites Reinfusion Therapy (CART).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2026-11-01 (Estimated); Primary Completion 2028-11-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | 12 months
  The overall response rate (ORR) of participants with an Eastern Cooperative Oncology Group performance status (PS) of 2 who receive single-agent trastuzumab deruxtecan as determined by the treating investigator using RECIST 1.1.

SECONDARY OUTCOMES:
Percentage of Study Participants with Toxic Side Effects in Response to Trastuzumab Deruxtecan | 12 months
  Percentage of subjects with treatment-emergent grade 3-4 toxicities, defined by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Overall Survival | 12 months
  Overall survival defined as the time from Day 1 of administering trastuzumab deruxtecan (Enhertu) to death from any cause.
Progression Free Survival | 12 months
  Progression free survival defined as the time from Day 1 of administering trastuzumab deruxtecan (Enhertu) until the criteria for disease progression is met as determined by the treating investigator using RECIST 1.1 or death as a result of any cause.
Disease Control Rate | 12 months
  Disease control rate defined as the proportion of participants with RECIST 1.1-based progressive disease, complete response and stable disease divided by the total number of evaluable participants.
Duration of Response | 12 months
  Duration of response defined as the time from disease response to progression or death. This will only calculated for the participants with response.

CONTACTS AND LOCATIONS:
Overall Officials: Manik Amin, MD, Principal Investigator — University of Chicago

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Loren AW, Mangu PB, Beck LN, Brennan L, Magdalinski AJ, Partridge AH, Quinn G, Wallace WH, Oktay K; American Society of Clinical Oncology. Fertility preservation for patients with cancer: American Society of Clinical Oncology clinical practice guideline update. J Clin Oncol. 2013 Jul 1;31(19):2500-10. doi: 10.1200/JCO.2013.49.2678. Epub 2013 May 28. PMID 23715580
- [Background] Garland SN, Pelletier G, Lawe A, Biagioni BJ, Easaw J, Eliasziw M, Cella D, Bathe OF. Prospective evaluation of the reliability, validity, and minimally important difference of the functional assessment of cancer therapy-gastric (FACT-Ga) quality-of-life instrument. Cancer. 2011 Mar 15;117(6):1302-12. doi: 10.1002/cncr.25556. Epub 2010 Oct 19. PMID 20960518
- [Background] Boku N, Yamamoto S, Fukuda H, Shirao K, Doi T, Sawaki A, Koizumi W, Saito H, Yamaguchi K, Takiuchi H, Nasu J, Ohtsu A; Gastrointestinal Oncology Study Group of the Japan Clinical Oncology Group. Fluorouracil versus combination of irinotecan plus cisplatin versus S-1 in metastatic gastric cancer: a randomised phase 3 study. Lancet Oncol. 2009 Nov;10(11):1063-9. doi: 10.1016/S1470-2045(09)70259-1. Epub 2009 Oct 7. PMID 19818685
- [Background] Enzinger PC, Kulke MH, Clark JW, Ryan DP, Kim H, Earle CC, Vincitore MM, Michelini AL, Mayer RJ, Fuchs CS. A phase II trial of irinotecan in patients with previously untreated advanced esophageal and gastric adenocarcinoma. Dig Dis Sci. 2005 Dec;50(12):2218-23. doi: 10.1007/s10620-005-3038-2. PMID 16416165
- [Background] Einzig AI, Neuberg D, Remick SC, Karp DD, O'Dwyer PJ, Stewart JA, Benson AB 3rd. Phase II trial of docetaxel (Taxotere) in patients with adenocarcinoma of the upper gastrointestinal tract previously untreated with cytotoxic chemotherapy: the Eastern Cooperative Oncology Group (ECOG) results of protocol E1293. Med Oncol. 1996 Jun;13(2):87-93. doi: 10.1007/BF02993858. PMID 9013471
- [Background] Ilson DH, Wadleigh RG, Leichman LP, Kelsen DP. Paclitaxel given by a weekly 1-h infusion in advanced esophageal cancer. Ann Oncol. 2007 May;18(5):898-902. doi: 10.1093/annonc/mdm004. Epub 2007 Mar 9. PMID 17351256
- [Background] Hall PS, Swinson D, Cairns DA, Waters JS, Petty R, Allmark C, Ruddock S, Falk S, Wadsley J, Roy R, Tillett T, Nicoll J, Cummins S, Mano J, Grumett S, Stokes Z, Kamposioras KV, Chatterjee A, Garcia A, Waddell T, Guptal K, Maisey N, Khan M, Dent J, Lord S, Crossley A, Katona E, Marshall H, Grabsch HI, Velikova G, Ow PL, Handforth C, Howard H, Seymour MT; GO2 Trial Investigators. Efficacy of Reduced-Intensity Chemotherapy With Oxaliplatin and Capecitabine on Quality of Life and Cancer Control Among Older and Frail Patients With Advanced Gastroesophageal Cancer: The GO2 Phase 3 Randomized Clinical Trial. JAMA Oncol. 2021 Jun 1;7(6):869-877. doi: 10.1001/jamaoncol.2021.0848. PMID 33983395
- [Background] Oken MM, Creech RH, Tormey DC, Horton J, Davis TE, McFadden ET, Carbone PP. Toxicity and response criteria of the Eastern Cooperative Oncology Group. Am J Clin Oncol. 1982 Dec;5(6):649-55. No abstract available. PMID 7165009
- [Background] Bang YJ, Van Cutsem E, Feyereislova A, Chung HC, Shen L, Sawaki A, Lordick F, Ohtsu A, Omuro Y, Satoh T, Aprile G, Kulikov E, Hill J, Lehle M, Ruschoff J, Kang YK; ToGA Trial Investigators. Trastuzumab in combination with chemotherapy versus chemotherapy alone for treatment of HER2-positive advanced gastric or gastro-oesophageal junction cancer (ToGA): a phase 3, open-label, randomised controlled trial. Lancet. 2010 Aug 28;376(9742):687-97. doi: 10.1016/S0140-6736(10)61121-X. Epub 2010 Aug 19. PMID 20728210
- [Background] Siegel RL, Miller KD, Fuchs HE, Jemal A. Cancer statistics, 2022. CA Cancer J Clin. 2022 Jan;72(1):7-33. doi: 10.3322/caac.21708. Epub 2022 Jan 12. PMID 35020204
- [Background] Torre LA, Siegel RL, Ward EM, Jemal A. Global Cancer Incidence and Mortality Rates and Trends--An Update. Cancer Epidemiol Biomarkers Prev. 2016 Jan;25(1):16-27. doi: 10.1158/1055-9965.EPI-15-0578. Epub 2015 Dec 14. PMID 26667886
- [Background] Sitarz R, Skierucha M, Mielko J, Offerhaus GJA, Maciejewski R, Polkowski WP. Gastric cancer: epidemiology, prevention, classification, and treatment. Cancer Manag Res. 2018 Feb 7;10:239-248. doi: 10.2147/CMAR.S149619. eCollection 2018. PMID 29445300